CLINICAL TRIAL: NCT03845842
Title: Randomized Controlled Trial of a Volitional Help Sheet in Cannabis Users
Brief Title: Using Implementation Intentions to Reduce Cannabis Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Lynsey Gregg, Principal Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018 5701
Record Dates: First submitted 2018-12-20; First posted 2019-02-19 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Cannabis Use
Keywords: Cannabis; Risk reduction
MeSH Terms: conditions — Marijuana Abuse; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (volitional help sheet) (Active Comparator): Participants read a brief statement designed to encourage them to reduce their cannabis use ("We want you to plan to reduce your cannabis use"). Participants are presented with a table with two columns and twenty rows. Twenty 'high risk' situations (temptations) are presented in the left hand column and 20 appropriate responses (processes of change) are presented in the right hand column (see Armitage, 2008). Participants are told that identifying situations in which they were tempted to use cannabis and identifying ways to overcome those temptations had been shown to help people change their behaviour and are asked to tick critical situations/appropriate responses that might be useful to them.
  Interventions: Behavioral: Volitional help sheet
- Intervention (volitional help sheet) (Experimental): Participants read a brief statement designed to encourage them to reduce their cannabis use ("We want you to plan to reduce your cannabis use"). Participants are presented with a table with two columns and twenty rows. Twenty 'high risk' situations (temptations) are presented in the left hand column and 20 appropriate responses (processes of change) are presented in the right hand column (see Armitage, 2008). Participants are told that identifying situations in which they were tempted to use cannabis and identifying ways to overcome those temptations had been shown to help people change their behaviour. Implementation intentions are formed by linking critical situations with appropriate responses by choosing an appropriate response from a drop down menu for each critical situation.
  Interventions: Behavioral: Volitional help sheet

INTERVENTIONS:
Behavioral: Volitional help sheet — Participants are asked to choose from a list of strategies for avoiding cannabis use.

SUMMARY:
The study will recruit frequent users of cannabis (defined at least fortnightly use) and randomize them either to: (1) form implementation intentions by linking situations in which they are tempted to use cannabis with strategies to avoid using cannabis in those situations by using a volitional help sheet, or (2) to consider the situations in which they are tempted to use cannabis alongside possible strategies to avoid using it as presented in the volitional help sheet but not to form implementation intentions. The effects on self-reported cannabis use will be assessed 1 month post-intervention. Predictors of cannabis reduction will also be examined.

DETAILED DESCRIPTION:
Design: This study will use questionnaires to assess participants cannabis habits (frequency and amount of use) and then employ planning strategies to help them quit. Follow up questionnaires will be used to ascertain the success of planning on reduction in cannabis use.

Sample Size: We plan to recruit a minimum of 60 participants in each condition (120 total) but aim to collect data from as many participants as possible.

Recruitment: To participate in this study a person must be over the age of 18 and a frequent user of cannabis. The study will be advertised online on social media platforms.

Procedure: Potential participants will follow an online link to a briefing sheet that provides information about the study. The sheet will also inform participants that they do not have to complete the questionnaire and that they can withdraw from the study at any time without giving a reason. Once they have read the briefing sheet and generated their personal identity code, as instructed, they will complete the questionnaire online. A month after the participants have completed the initial questionnaire they will receive a link to a follow-up questionnaire via email. Email addresses will be stored separately to study data and will be destroyed once the follow up phase has completed and their involvement in the study ends.

Outcomes and Analysis: The main purpose of this study is to explore the role of planning in encouraging people to reduce cannabis use. Quantitative analysis will be conducted to assess the effects of planning on cannabis use reduction. The investigators expect to find that planning is effective in helping people reduce their use.

ELIGIBILITY:
Inclusion Criteria:

* Frequent cannabis user (at least fortnightly)

Exclusion Criteria:

* Younger than 18 years of age
* Infrequent / no cannabis use (less than fortnightly)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Cannabis use reduction (amount) | 1 month
  Self-reported cannabis use -amount of cannabis (weight)
Cannabis use reduction (frequency) | 1 month
  Self-reported cannabis use - frequency of use (days per week)

SECONDARY OUTCOMES:
Self reported habit as measured by the automaticity subscale of the Self-Report Habit Index. | 1 month
  Self-reported habit (e.g., "Using cannabis is something I do automatically: strongly agree - strongly disagree).
Self reported action control as measured by the scale developed by Sniehotta et al (2011) | 1 month
  Self-reported action control (e.g., "During the last week I often had my intention to reduce my cannabis use on my mind: strongly disagree-strongly agree")
Self reported craving as measured by items from the mood and physical symptoms scale (MPSS) | 1 month
  self reported craving

CONTACTS AND LOCATIONS:
Overall Officials: Lynsey Gregg, PhD, Principal Investigator — The University of Manchester
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sniehotta FF, Nagy G, Scholz U, Schwarzer R. The role of action control in implementing intentions during the first weeks of behaviour change. Br J Soc Psychol. 2006 Mar;45(Pt 1):87-106. doi: 10.1348/014466605X62460. PMID 16573874
- [Background] Gardner B, Abraham C, Lally P, de Bruijn GJ. Towards parsimony in habit measurement: testing the convergent and predictive validity of an automaticity subscale of the Self-Report Habit Index. Int J Behav Nutr Phys Act. 2012 Aug 30;9:102. doi: 10.1186/1479-5868-9-102. PMID 22935297
- [Background] West R, Hajek P. Evaluation of the mood and physical symptoms scale (MPSS) to assess cigarette withdrawal. Psychopharmacology (Berl). 2004 Dec;177(1-2):195-9. doi: 10.1007/s00213-004-1923-6. Epub 2004 Jun 4. PMID 15179542